CLINICAL TRIAL: NCT02979548
Title: Study to Evaluate the Anti-emetic Effect of Aprepitant as an add-on Therapy in Children and Adolescents Receiving AML Remission Induction Chemotherapy: An Investigator-initiated, Randomized, Open Label Trial
Brief Title: Study to Evaluate the Effect of Aprepitant in Children and Adolescents Receiving AML Remission Induction Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Atul Sharma (Other)
Responsible Party: Sponsor-Investigator, Dr Atul Sharma, Senior Resident, All India Institute of Medical Sciences
Organization: All India Institute of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IECPG-419
Record Dates: First submitted 2016-11-28; First posted 2016-12-01 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Chemotherapy Induced Vomiting; Acute Myeloid Leukemia
Keywords: Aprepitant
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Aprepitant; Ondansetron; Metoclopramide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A : Aprepitant (Add on therapy) (Experimental): Aprepitant group will receive aprepitant capsules 1 h prior to chemotherapy on days 1-3 in addition to 5HT3 RA (Ondansetron). The dose of aprepitant will be given based on weight groups Weight 15-40 kg : Aprepitant 80 mg on days 1-3 Weight > 41kg: Aprepitant 125 mg on day 1 followed by 80 mg on days 2-3 Rescue medication, injection metoclopramide 0.5 mg/kg body weight/day.
  Interventions: Drug: Aprepitant; Drug: Ondansetron; Drug: Metoclopramide
- Group B : 5HT3 RA (Ondansetron) (Active Comparator): On the day of chemotherapy, ondansetron will be administered to all patients as per our institutional practice in a dose of 0.15 mg/kg as an intravenous bolus 30 minutes before chemotherapy followed by every 8 hourly for 8 days.
  Rescue medication, injection metoclopramide 0.5 mg/kg body weight/day.
  Interventions: Drug: Ondansetron; Drug: Metoclopramide

INTERVENTIONS:
Drug: Aprepitant — Aprepitant is a non peptide, selective, Neurokinin type 1 (NK 1) receptor antagonist. Group A will receive Aprepitant as an add-on anti-emetic therapy in addition to ondansetron.
  Other Names: Apretero
  Arms: Group A : Aprepitant (Add on therapy)
Drug: Ondansetron — Ondansetron is 5HT3 Receptor antagonist used to treat and prevent chemotherapy induced nausea and vomiting
  Other Names: Zofer, Emset
Drug: Metoclopramide — Dopamine receptor antagonist , acts at CTZ. Rescue medication, injection metoclopramide 0.5 mg/kg body weight/day.
  Other Names: Reglan

SUMMARY:
The purpose of the study is to find out the efficacy of an anti-emetic drug, Aprepitant as an add-on therapy to prevent vomiting in children and adolescents receiving chemotherapy for leukemia (AML).

Children and adolescents admitted with confirmed diagnosis of AML will be assessed for eligibility criteria and enrolled in the study. Then they will be divided (randomized) into experimental and control groups.

Experimental group will receive Aprepitant capsules 1 h prior to chemotherapy on days 1-3 in addition to ondansetron. Patients will be required to swallow the whole capsule and opening of capsule will not be permitted. All three doses will be administered under supervision.

Control group will receive ondansetron (0.15 mg/kg) as an intravenous bolus 30 minutes before chemotherapy followed by every 8 hourly for 8 days. Metoclopramide will be used as a rescue agent.

The data will be collected from each patient in a proforma from day 1 to day 13 of chemotherapy. A Diary will be maintained for nausea and vomiting record.

Edmonton's symptom assessment criterion will be used in the diary for assessing severity of nausea. The NCI guidelines will be used to assess the severity of vomiting based on the data provided by the patient in the diary.

A modified intention-to-treat population (patients who receive chemotherapy, take one or more doses of study drug, and have one or more post treatment measurements) will be used for efficacy analysis. Proportion of patients with complete response will be compared between patients with or without aprepitant.

DETAILED DESCRIPTION:
Children and adolescents admitted with confirmed diagnosis of AML will be assessed for eligibility criteria and enrolled in the study. Subjects will be randomized into experimental and control groups using table of random numbers generated by computer.Experimental group will receive aprepitant capsules as an add-on therapy (Apretero; Hetero Laboratories, India) 1 h prior to chemotherapy on days 1-3 in addition to ondansetron.

The dose of aprepitant will be as per our previous study based on weight groups'

* Weight 15-40 kg : Aprepitant 80 mg on days 1-3
* Weight > 41kg: Aprepitant 125 mg on day 1 followed by 80 mg on days 2-3 Patients will be required to swallow the whole capsule and opening of capsule will not be permitted.

All three doses will be administered under supervision by the sister allocated. Control group will receive ondansetron (0.15 mg/kg) as an intravenous bolus 30 minutes before chemotherapy followed by every 8 hourly. Metoclopramide will be used as a rescue agent.

The data will be collected from each patient in a proforma from day 1 to day 13 of chemotherapy by the investigator during his/her stay as in-patient in the hospital. The Proforma will contain different items dealing with demographic and clinical characteristic of the subjects.A Diary will be maintained for nausea and vomiting record. It will help in collecting data regarding nausea, vomiting along with some additional variables like- chemotherapy related toxicities, requirement of any rescue medication.

The subjects will be given the diary for symptom assessment on day 1 and it will be filled up under the supervision of the investigator on day 1 and day 2 of chemotherapy. The diary will be given to the subjects on day 3 of the chemotherapy to record all the events (incidence and severity of nausea, vomiting, requirement of rescue medication and other toxicities).

Edmonton's symptom assessment criterion will be used in the diary for assessing severity of nausea. The NCI guidelines will be used to assess the severity of vomiting based on the data provided by the patient in the diary.Patients/attendant's will be explained about the filling of the diary and will maintain it for recording of vomiting under the investigator's supervision.

A modified intention-to-treat population (patients who receive chemotherapy, take one or more doses of study drug, and have one or more post treatment measurements) will be used for efficacy analysis.Proportion of patients with CR will be compared between patients with or without aprepitant.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, chemotherapy-naïve de novo AML patients planned for 3+7 remission induction chemotherapy in the age group 5-18 years
2. Weight above 15 kg (Those who are able to swallow the medication )
3. Children/adolescents and their caregiver who can understand Hindi or English and willing to participate in the study (with written informed consent)

Exclusion Criteria:

1. Vomiting/retching within 24 h prior to treatment
2. Significant organ dysfunction (aspartate aminotransferase/alanine aminotransferase >2.5 times of upper normal limit, serum bilirubin >1.5 times of upper normal limit, serum creatinine>1.5 times of upper normal limit)
3. Patient on inotropic support at presentation
4. Patient with respiratory failure/mechanical ventilation at presentation

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with complete response during the acute phase of AML remission induction chemotherapy | Up to day 8 of induction

SECONDARY OUTCOMES:
Time to first episode of vomiting | Up to day 13
Incidence of delayed vomiting | From day 9 to day 13
Severity of vomiting | Up to day 13
  Severity will be assessed by NCI CTCAE Criteria version 4.0
Incidence of requirement of rescue medication | Up to day 8

CONTACTS AND LOCATIONS:
Locations (1):
- Irch, Aiims , New Delhi , India, New Delhi, DEL, India

IPD SHARING:
Plan to Share IPD: Undecided
It is undecided but if required the data can be made available.

REFERENCES:
- [Derived] Sharma A, Ganguly S, C SK, Pillai AS, Dhawan D, Sreenivas V, Bakhshi S. Addition of aprepitant improves acute emesis control in children and adolescents receiving induction chemotherapy for acute myeloid leukaemia: a randomised, open-label trial. BMJ Support Palliat Care. 2023 Oct;13(e1):e156-e162. doi: 10.1136/bmjspcare-2020-002595. Epub 2020 Oct 29. PMID 33122168